CLINICAL TRIAL: NCT03266393
Title: A Prospective, Randomized, Single-center, Pilot Study of Envarsus XR® to Examine Safety, Medication Adherence, and Patient Reported Outcomes in Adolescent Renal Transplant Recipients
Brief Title: Envarsus XR® in Adolescent Renal Transplant Recipients
Acronym: EnvarsusXR
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Rachana Srivastava, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17-006138
Record Dates: First submitted 2017-08-10; First posted 2017-08-30 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Kidney Transplantation; Renal Transplantation; Grafting, Kidney
Keywords: Envarsus XR; Kidney transplantation; Grafting, Kidney; Tacrolimus; Rejection; Adherence; Quality of Life; post-transplant immunosuppression
MeSH Terms: conditions — Rejection, Psychology | interventions — Tacrolimus

STUDY DESIGN:
Intervention Model Description: Once enrolled, patients will be randomized 1:1 to immediate release tacrolimus that the patient had been maintained on prior to the study (twice daily formulation) or Envarsus XR® using a permuted block randomization sequence to improve the likelihood of balance between groups. Following randomization, and independent of the formulation of tacrolimus, each patient will have a "run-in" period of 14 days to optimize the dose to reach a tacrolimus trough level within their therapeutic target. Randomization will be stratified based on each patient's follow-up period post-transplant in 2 stratification groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A-Tacrolimus then Envarsus (Experimental): Immediate release tacrolimus (twice a day oral formulation) 14 day run-in followed by 4 months of follow-up and then crossing over to Envarsus XR® with a 14 day run-in followed by 4 months of follow-up.
  Interventions: Drug: Envarsus XR; Drug: Tacrolimus
- Arm B-Envarsus then Tacrolimus (Experimental): Envarsus XR® 14 day run-in followed by 4 months of follow-up and then crossing over to immediate release tacrolimus (twice a day oral formulation) with a 14 day run-in followed by 4 months of follow-up.
  Interventions: Drug: Envarsus XR; Drug: Tacrolimus

INTERVENTIONS:
Drug: Envarsus XR — Once daily sustained-release tacrolimus
  Other Names: extended release tacrolimus
Drug: Tacrolimus — Twice daily immediate-release tacrolimus
  Other Names: immediate release tacrolimus

SUMMARY:
Adolescents commonly experience barriers to adherence that entail forgetfulness, distraction, poor planning, and scheduling problems. A once daily oral regimen may be superior to the current regimens that require twice daily dosing. It is currently unclear if Envarsus XR® would improve outcomes in adolescent organ transplant recipients. Each patient will receive tacrolimus (twice daily immediate release oral formulation) which they are using as part of their standard of care immunosuppressive regimen for a portion of the study and Envarsus XR® (a once daily extended-release oral tacrolimus formulation) for a portion of the study in a cross-over design. Besides the advantage to adherence behaviors, a sustained-release tacrolimus preparation may decrease burdensome side effects and increase quality of life. Following enrollment, each patient will be maintained in the study for 9 months.

DETAILED DESCRIPTION:
This is a randomized, prospective, single-center, pilot study assessing once daily Envarsus XR® medication efficacy, adverse events, medication non-adherence, patient-reported outcomes, and abbreviated pharmacokinetics/ dose finding to evaluate a population of adolescent renal transplant recipients while on stable tacrolimus (twice daily) and then after conversion to Envarsus XR® to provide critical efficacy, safety, dose-finding, adherence, and patient reported outcome data that could lead to adoption of Envarsus XR® as a mainstay of pediatric/adolescent post-transplant immunosuppression.

Following randomization, and independent of the formulation of tacrolimus, each patient will have a "run-in" period of 14 days to optimize the dose to reach a tacrolimus trough level of 4 to 10 ng/ml.

* Drug Administration: After randomization (to either twice daily tacrolimus or once daily Envarsus ®) and the "run-in" period, patients will be continued on their assigned tacrolimus formulation for 4 months. He/she will then be then switched to the opposite tacrolimus formulation. Following the switch, there will be a 14 day run-in period to establish the optimal trough level (4-10 ng/ml) (analogous to the first run-in period) and then continued on that tacrolimus formulation for 4 months.
* Pharmacokinetics: Irrespective of whether a patient starts on Envarsus XR® after randomization or is switched to Envarsus XR® after 4 months of immediate release tacrolimus, the dose of Envarsus XR® will be determined by using a dose conversion ratio targeting 0.7 (but may range from 0.66-0.8 because of dosage strengths of Envarsus XR® dosing formulations) relative to the immediate release formulation that he/she was receiving as maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of first kidney transplants (deceased or living donor) with stable allograft function
* 6 or more months after transplantation
* Currently on a stable dose of twice-daily tacrolimus and mycophenolate mofetil (MMF) or enteric coated mycophenolic acid (EC-MPA)± corticosteroids for a minimum of 6 months prior (patient has remained on a dosing that has changed no greater than ± 0.5mg/dose for a minimum of 4 months)
* Ability to comply with study procedures for the entire length of the study
* Patient and/or parent/legal guardian has been informed about the study survey and has signed an informed consent form.

Exclusion Criteria:

* Detectable donor specific anti-HLA antibody prior to enrollment (pre- or post-transplant)
* Actively being treated for an episode of biopsy proven acute cellular rejection (ACR) (Banff 1A or greater)
* Post-transplant history of biopsy proven ACR (Banff 1B or greater) or antibody mediated rejection (AMR)
* Currently receiving, planning to receive, or received within 7 days prior to study enrollment any drug interacting or interfering with tacrolimus metabolism (azole antifungals, erythromycin, clarithromycin, diltiazem, protease inhibitors, statins, grapefruit juice, rifampin or anti-seizure medications shown to interact with tacrolimus)
* Currently receiving an mTOR inhibitor (sirolimus, everolimus)
* Gastrointestinal illness that might affect the absorption of tacrolimus
* Unable or unwilling to complete study survey questionnaire
* Professional care taker is responsible for dispensing subject's medication
* Recipient of HLA identical or zero HLA mismatched organ transplant
* Documented history of medication non-adherence following transplantation prior to enrollment

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of clinical or subclinical allograft injury at any timepoint as assessed by the appearance of de novo donor specific anti-HLA antibody (dnDSA) OR biopsy proven allograft rejection. | 9 months
  Appearance of dnDSA will be assessed by Luminex Single Antigen Bead assay. Patients will be monitored for rejection by measuring serum creatinine, a marker of renal function. If the creatinine level suggests allograft dysfunction, a biopsy will be performed and the tissue assessed by the 2013 Banff Criteria to determine presence of absence of rejection. Incidence rates will be compared across 4 month follow-up periods of each for twice-daily tacrolimus and Envarsus XR® descriptively and using Poisson or negative binomial models with random coefficients (intercepts or slopes) to account for nesting of assessment time points within individuals.
Change in Patient Reported Transplant Symptoms | Baseline, 2.5 months, 4.5 months, 7 months, 9 months
  Change in transplant symptoms will be assessed longitudinally by the Modified Transplant Symptom Occurrence and Distress Scale (MTSODS-59R). The MTSODS-59R assesses 59 side effects from immunosuppressive medications. Scores on each measure will be calculated and described with means, medians, standard deviations, and ranges. Change within individuals will be summarized descriptively, plotted over the study timepoints, and analyzed with repeated measures random coefficients models (unconditional model with no predictors). These models will determine if there is a significant difference in these outcomes when patients are on twice-daily tacrolimus and Envarsus XR®.
Change in Patient Reported Medication Adherence and Barriers | Baseline, 2.5 months, 4.5 months, 7 months, 9 months
  Outcome will be assessed longitudinally by the Basel Assessment of Adherence with Immunosuppressive Medication Scale (BASIS), Adolescent and Parent Medication Barriers Scale (AMBS/PMBS), and Attitudes Toward Transplant Scale - Patient (ATTS-P). The BASIS assesses adherence in the last 4 weeks (did not take dose, forgetting dose, perception of not needing, reducing amount). The AMBS/PMBS are 17/16 item scales measuring medication barriers (Disease Frustration/Adolescent Issues, Ingestion Issues, Regimen Adaptation/Cognitive). The ATTS-P 4 item "Attitudes toward Medication" subscale (e.g., "Medication is not a problem - problematic, "Medication is a relief - burdensome") will also be used. Scores on each measure will be calculated and numerically described. Change within individuals will be summarized descriptively, plotted over the study timepoints, and analyzed with repeated measures random coefficients models (unconditional model with no predictors) comparing mediation regimens.
Incidence of Adverse Events (AE) and Serious Adverse Events (SAE) as a measure of safety | 2 weeks, 2.5 months, 4.5 months, 5 months, 7 months, 9 months
  Patients will be monitored for for the appearance of AEs or SAEs. Rates will be compared across 4 month follow-up periods of each for twice-daily tacrolimus and Envarsus XR® descriptively and using Poisson or negative binomial models with random coefficients (intercepts or slopes) to account for nesting of assessment time points within individuals.
Change in Patient Reported Distress | Baseline, 2.5 months, 4.5 months, 7 months, 9 months
  Change in distress will be assessed longitudinally by the Patient Reported Outcomes Measurement Information System (PROMIS®) Pediatric/Parent Proxy Profile 25. The PROMIS® includes 25 questions generating several subscales for fatigue, pain interference, pain intensity, physical function-mobility, anxiety, depressive symptoms, and peer relationships. Scores on each measure will be calculated and described with means, medians, standard deviations, and ranges. Change within individuals will be summarized descriptively, plotted over the study timepoints, and analyzed with repeated measures random coefficients models (unconditional model with no predictors). These models will determine if there is a significant difference in these outcomes when patients are on twice-daily tacrolimus and Envarsus XR®.

SECONDARY OUTCOMES:
Tacrolimus Dose Exposure | Day 14 after starting Envarsus XR ®
  Measured as area-under the curve (AUC), based on a limited sampling strategy. On day 14 after starting Envarsus XR ® patients will have an abbreviated pharmacokinetic assessment using the following time points: 0 hours (trough pre-dose) and at 8 and 12 hours post-dose. The AUC will be described.
Tacrolimus Trough Coefficient of Variation | Baseline; Days 7, 14, 44, 74, 104, 134, 142, 148, 178, 208, 238, 268
  To determine the association between tacrolimus trough level % coefficient of variation (CV%) and patient non-adherence self- reporting and compare these measures between twice daily tacrolimus and Envarsus XR®. CV% will be calculated as CV% = (standard deviation/mean) × 100 of tacrolimus trough levels collected while taking each tacrolimus formulation.
Incidence of IgG3 and C1q positive Donor Specific Antibodies | Baseline, 2.5 months, 4.5 months, 7 months, 9 months
  To determine the association of non-adherence with the development of IgG3 and C1q positive dnDSA. Incidence rates will be compared across 4 month follow-up periods of each for twice-daily tacrolimus and Envarsus XR® descriptively and using Poisson or negative binomial models with random coefficients (intercepts or slopes) to account for nesting of assessment time points within individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Rachana Srivastava, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Transplantation Services, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Filler G, Grygas R, Mai I, Stolpe HJ, Greiner C, Bauer S, Ehrich JH. Pharmacokinetics of tacrolimus (FK 506) in children and adolescents with renal transplants. Nephrol Dial Transplant. 1997 Aug;12(8):1668-71. doi: 10.1093/ndt/12.8.1668. PMID 9269646
- [Background] Min SI, Ha J, Kang HG, Ahn S, Park T, Park DD, Kim SM, Hong HJ, Min SK, Ha IS, Kim SJ. Conversion of twice-daily tacrolimus to once-daily tacrolimus formulation in stable pediatric kidney transplant recipients: pharmacokinetics and efficacy. Am J Transplant. 2013 Aug;13(8):2191-7. doi: 10.1111/ajt.12274. Epub 2013 Jun 4. PMID 23734831
- [Background] Rostaing L, Bunnapradist S, Grinyo JM, Ciechanowski K, Denny JE, Silva HT Jr, Budde K; Envarsus Study Group. Novel Once-Daily Extended-Release Tacrolimus Versus Twice-Daily Tacrolimus in De Novo Kidney Transplant Recipients: Two-Year Results of Phase 3, Double-Blind, Randomized Trial. Am J Kidney Dis. 2016 Apr;67(4):648-59. doi: 10.1053/j.ajkd.2015.10.024. Epub 2015 Dec 22. PMID 26717860
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829